CLINICAL TRIAL: NCT02213263
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND STUDY OF PF-05280586 VERSUS RITUXIMAB FOR THE FIRST-LINE TREATMENT OF PATIENTS WITH CD20-POSITIVE, LOW TUMOR BURDEN, FOLLICULAR LYMPHOMA
Brief Title: A Study Of PF-05280586 (Rituximab-Pfizer) Or MabThera® (Rituximab-EU) For The First-Line Treatment Of Patients With CD20-Positive, Low Tumor Burden, Follicular Lymphoma (REFLECTIONS B328-06)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B3281006; 2014-000132-41 (EudraCT Number); REFLECTIONS (Other: Alias Study Number)
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Follicular Lymphoma
Keywords: rituximab; follicular lymphoma; Non-Hodgkin lymphoma; Non-Hodgkin's lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Non-Hodgkin | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF-05280586 (Experimental)
  Interventions: Biological: PF-05280586
- MabThera® (Active Comparator)
  Interventions: Biological: MabThera®

INTERVENTIONS:
Biological: PF-05280586 — PF-05280586 (rituximab-Pfizer) concentrate for solution for infusion 375mg/m2 administered via IV infusion on Days 1, 8, 15, and 22
  Arms: PF-05280586
Biological: MabThera® — MabThera® (rituximab-EU) concentrate for solution for infusion 375mg/m2 administered via IV infusion on Days 1, 8, 15, and 22
  Arms: MabThera®

SUMMARY:
This study will compare the safety and effectiveness of PF-05280586 versus rituximab-EU in patients with CD20-positive, low tumor burden follicular lymphoma. The primary hypothesis to be tested in this study is that the effectiveness of PF-05280586, as measured by the Overall Response Rate, is similar to that of rituximab-EU.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of low tumor burden, CD20-positive follicular lymphoma
* Ann Arbor Stage II, III, or IV

Exclusion Criteria:

* Not a candidate for treatment with rituximab as a single-agent
* Evidence of transformation to a high grade or diffuse large B-cell lymphoma
* Any previous systemic therapy for B-cell NHL, including chemotherapy, immunotherapy, or steroids
* Any prior treatment with rituximab
* Active, uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2018-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (413):
- United States (84):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - The Oncology Institute of Hope and Innovation, Anaheim, California
  - Compassionate Care Research Group, Inc., at Compassionate Cancer Care Medical Group, Inc., Corona, California
  - The Oncology Institute of Hope and Innovation, Downey, California
  - Compassionate Care Research Group, Inc., at Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Global Cancer Research Institute (GCRI), Inc, Gilroy, California
  - Saint Louise Regional Hospital Radiology Department (Radiology Only), Gilroy, California
  - South Valley Imaging Center (Imaging Only), Gilroy, California
  - Los Angeles Hematology Oncology Medical Group, Glendale, California
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - The Oncology Institute of Hope and Innovation, Long Beach, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - The Oncology Institute of Hope and Innovation, Lynwood, California
  - The Oncology Institute of Hope and Innovation, Montebello, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - Torrance Health Association DBA, Torrance Memorial Physician, Network/Cancer Care Associates, Redondo Beach, California
  - Compassionate Care Research Group, Inc., at Compassionate Cancer Care Medical Group, Inc., Riverside, California
  - Global Cancer Research Institute, Inc., San Jose, California
  - O'Connor Hospital, San Jose, California
  - PET Imaging of San Jose (Imaging Only), San Jose, California
  - The Oncology Institute of Hope and Innovation, Santa Ana, California
  - Torrance Memorial Medical Center, Torrance, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Innovative Clinical Research Institute (ICRI), Whittier, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Center-Lakewood (Laboratory), Lakewood, Colorado
  - Rocky Mountain Cancer Centers (RMCC) - Lakewood - St Anthony, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Center Pueblo, Pueblo, Colorado
  - John D. Archbold Memorial Hospital, Thomasville, Georgia
  - Lewis Hall Singletary Oncology Center At John D. Archbold Memorial Hospital, Thomasville, Georgia
  - Northwestern Medicine West Region, DeKalb, Illinois
  - Cancer Center,Northwestern Medicine, West Region, Geneva, Illinois
  - Cancer Center of Kansas, Chanute, Kansas
  - Cancer Center of Kansas, Dodge City, Kansas
  - Cancer Center of Kansas, El Dorado, Kansas
  - Cancer Center of Kansas, Independence, Kansas
  - Cancer Center of Kansas, Kingman, Kansas
  - Cancer Center of Kansas, Liberal, Kansas
  - Cancer Center of Kansas, McPherson, Kansas
  - Cancer Center of Kansas, Newton, Kansas
  - The University of Kansas Cancer Center, Overland Park, Kansas
  - Cancer Center of Kansas, Parsons, Kansas
  - Cancer Center of Kansas, Salina, Kansas
  - Cancer Center of Kansas, Wellington, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Cancer Center Of Kansas, Winfield, Kansas
  - PET/CT facility Seton Imaging Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Rcca Md Llc, Bethesda, Maryland
  - Holy Cross Hospital Resource Center, Silver Spring, Maryland
  - Holy Cross Hospital Hospital Pharmacy, Silver Spring, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Maryland Oncology Hematology, P.A., Wheaton, Maryland
  - The University of Kansas Cancer Center, Kansas City, Missouri
  - The University of Kansas Cancer Center, Lee's Summit, Missouri
  - Saint Francis Medical Center, Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Saint Francis Medical Center, Grand Island, Nebraska
  - Saint Francis Medical Center, Saint Francis Cancer Treatment Center, Hastings, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Vidant Medical Center Pharmacy, Greenville, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Toledo Clinic Cancer Center - Maumee, Maumee, Ohio
  - Toledo Clinic Cancer Center - Toledo, Toledo, Ohio
  - Toledo Clinic, Inc., Toledo, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - San Antonio Military Medical Center- Department of Pharmacy, Fort Sam Houston, Texas
  - San Antonio Military Medical Center- Department of Radiology, Fort Sam Houston, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Investigational Products Center (I PC), Fort Worth, Texas
  - Investigational Products Center (IPC), Fort Worth, Texas
  - Millennium Oncology, Houston, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - Millennium Oncology, Kingwood, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Millennium Oncology, Shenandoah, Texas
  - Millennium Oncology, The Woodlands, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Yakima Valley Memorial Hospital/North Star Lodge Cancer Center, Yakima, Washington
- Austria (2):
  - Krankenhaus der Barmherzigen Schwestern Linz, Linz
  - Kepler Universitaetsklinikum GmbH, Linz
- Belarus (4):
  - SI 'Republican Research and Practice Centre of Oncology and Medical Radiology n.a. N.N. Alexandrov', Lyasny, Minsk Oblast
  - Healthcare Institution "Brest Regional Oncologic Dispensary", Brest
  - Healthcare Institution 'Minsk City Clinical Oncology Dispensary', Minsk
  - SI Republican Research and Practice Centre of oncology and medical radiology n.a N.N Alexandrov, Republic of Belarus
- Belgium (10):
  - Hopital Erasme, Brussels
  - Nuclear Medicine Department, Brussels
  - Grand Hopital de Charleroi-Site Notre-Dame, Charleroi
  - PET/CT facility: Grand Hopital de Charleroi (GHdC) - site Notre-Dame, Charleroi
  - Pharmacy Department: Grand Hopital de Charleroi (GHdC) - site Notre-Dame, Charleroi
  - Pharmacy Department, Centre Hospitalier De Jolimont - Lobbes, La Louviere (Haine-Saint Paul)
  - Centre Hospitalier de Jolimont - Lobbes, La Louviere (Haine-Saint-Paul)
  - Radiology Department, La Louviere (Haine-Saint-Paul)
  - C.H.U. Ambroise Pare, Mons
  - Pharmacy Department, CHU Ambroise Pare, Mons
- Brazil (30):
  - Hospital Santa Izabel - Setor de Bioimagem, Salvador, Estado de Bahia
  - Hospital Santa Izabel / Santa Casa de Misericordia da Bahia, Salvador, Estado de Bahia
  - Clinica Multimagem, Goiânia, Goiás
  - Hospital das Clinicas da Universidade Federal de Goias \ Centro de Pesquisa Clinica, Goiânia, Goiás
  - Centro de Imagens da Faculdade de Medicina - INCT Medicina Nuclear - PET/CT, Belo Horizonte, Minas Gerais
  - Hospital das Clinicas Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Unidade Funcional Apoio Diagnostico e terapeutica por Imagem do HC/UFMG - CT Scan, Belo Horizonte, Minas Gerais
  - Central de Misturas Intravenosas do Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre - Centro de Pesquisa Clinica, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Servico de Radiologia do Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - CDI - Centro de Diagnostico por Imagem do Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - InsCer - Instituto do Cerebro do Rio Grande do Sul - PUCRS, Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia (UBEA) - Hospital Sao Lucas da PUCRS -, Porto Alegre, Rio Grande do Sul
  - CEMEDI, Campinas, São Paulo
  - Instituto Radium, Campinas, São Paulo
  - CAEP - Centro Avancado de Estudos e Pesquisas LTDA, Campinas, São Paulo
  - Hospital e Maternidade Madre Theodora LTDA, Campinas, São Paulo
  - CENNI Oncologia, Campinas, São Paulo
  - Fundacao Amaral Carvalho / Fundacao Dr. Amaral Carvalho, Jaú, São Paulo
  - Unidade de Quimioterapia, Jaú, São Paulo
  - Casa da Esperanca, Santo André, São Paulo
  - Fundacao do ABC - FMABC/ Faculdade de Medicina ABC ( CEPHO - Centro de Estudos e Pesquisas de, Santo André, São Paulo
  - Tecnolab, São Bernardo do Campo, São Paulo
  - IEP São Lucas (Pharmacy), São Paulo, São Paulo
  - Hospital Bandeirantes, São Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da USP / Fundacao Faculdade de Medicina MEC MPAS, São Paulo, São Paulo
  - Casa de Saude Santa Marcelina (Centro de Pesquisa Santa Marcelina), São Paulo, São Paulo
  - IEP Sao Lucas - Instituto de Ensino e Pesquisa Sao Lucas / HEMOMED - Instituto de Oncologia e, São Paulo
  - Fleury, São Paulo
- Croatia (5):
  - University Hospital Center Zagreb, Department of Nuclear Medicine and Radiation Protection, Zagreb
  - University Hospital Center Zagreb, Department of Pathology and Cytology, Zagreb
  - University Hospital Center Zagreb, Department of Radiology, Zagreb
  - University Hospital Centre "Sestre Milosrdnice", Zagreb
  - University Hospital Centre Zagreb, Zagreb
- France (9):
  - CHU Marseille Hopital de La Conception, Marseille, Marseille Cedex 05
  - CH de Mulhouse, Hopital Emile Muller, Mulhouse, Mulhouse Cedex
  - Hopital Duchenne Chu - Boulogne Sur Mer, Boulogne-sur-Mer, NAP
  - Hopital Duchenne Chu - Boulogne Sur Mer, Boulogne-sur-Mer
  - Centre Hospitalier De Bourg En Bresse, Bourg-en-Bresse
  - Hopital Morvan-CHU Brest- Service Hematologie Clinique, Brest
  - Centre Hospitalier Universitaire Cote de Nacre, Caen
  - Centre Hospitalier du Mans, Le Mans
  - Clinique de la Sauvegarde, Lyon
- Georgia (3):
  - "LTD ""M. Zodelava's Hematology Centre""", Tbilisi
  - LTD "Research Institute of Clinical Medicine", Tbilisi
  - High Technology Medical Center, University Clinic, Tbilisi
- Germany (24):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Charite - Universitatsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charite - Universitaetsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - Charite - Universitatsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - Charite - Universitatsmedizin Berlin, Berlin
  - Klinikum Chemnitz gGmbH - Institut fuer Interventionelle Radiologie und Neuroradiologie, Chemnitz
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikum Chemnitz gGmbH - Klinik fuer Nuklearmedizin, Chemnitz
  - Klinikum Chemnitz gGmbH - Zentralapotheke, Chemnitz
  - Praxis im Koeln Triangle, Cologne
  - Universitaetsklinikum Essen (AoeR), Essen
  - Universitatsklinikum Essen (AoR), Essen
  - DokuSan Gesellschaft fuer Medizinische Studien mbH & Co. KG, Herne
  - Apotheke des St. Anna Hospital, Herne
  - EVK Eickel, Herne
  - Gemeinschaftspraxis fuer Diagnostische Radiologie und Nuklearmedizin, Mutlangen
  - Kliniken Ostalb, Stauferklinikum Schwaebisch Gmuend, Zentrum fuer Innere Medizin, Mutlangen
  - Stauferklinikum Schwaebisch Gmuend, Apotheke, Mutlangen
  - Universitaetsmedizin Rostock, Rostock
  - Klinikum Stuttgart, Klinik fuer Nuklearmedizin, Stuttgart
  - Vinzenz von Paul Kliniken gGmbH, Stuttgart
  - Radiologie Rhein-Sieg, Troisdorf
  - Ueberoertliche Berufsausuebungsgemeinschaft Drs. med. Helmut Forstbauer, Troisdorf
  - Zentralapotheke, Troisdorf
- Greece (12):
  - Gen. Hosp. of Athens "Evangelismos - Eye Hosp.- Polikliniki", Athens
  - Gen. Hosp. of Athens "Evangelismos-Eye Hosp. - Polikliniki", Athens
  - Gen. Hosp. of Athens "Evangelismos-Eye Hosp.-Polikliniki", Athens
  - Gen.Hosp.of Athens "Evangelismos-Eye Hosp.-polikiliniki", Athens
  - General Hospital of Athens "Evangelismos - Eye Hosp. - Polikliniki", Athens
  - Bioiatriki S.A., Athens
  - Bioiatriki, Athens
  - General Hospital of Athens 'Laiko', Athens
  - """ATTIKON"" Gen. Univ. Hosp", Athens
  - "ATTIKON'' Gen. Univ. Hosp., Chaidari, Athens
  - Magnitiki Patron, Pátrai
  - University General Hospital of Patras, Pátrai
- India (19):
  - Super Scan Imaging Centre, Surat, Gujarat
  - Pathology Department, Unique Hospital Multispeciality & Research Institute, Surat, Gujarat
  - Zircon- BIC Imaging Centre, Surat, Gujarat
  - HealthCare Global Enterprises Limited, Bangalore, Karnataka
  - Mangalore Institute of Oncology, Mangalore, Karnataka
  - Kasturba Medical College and Hospital, Manipal, Karnataka
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Department of Radiology, Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Department of Radiology, Pune, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - Ruby Hall clinic, Pune, Maharashtra
  - R.K. Birla Cancer Center, Sawai Man Singh Hospital, Jaipur, Rajasthan
  - Apollo Speciality Hospital, Chennai, Tamil Nadu
  - Department of Radiology, Chennai, Tamil Nadu
  - Global Hospitals, Hyderabad, Telangana
  - Vijaya Diagnostic Centre, Hyderabad, Telangana
  - N.R.S Medical College and Hospital, Kolkata, West Bengal
  - Spandan PET-CT Unit, Kolkata, West Bengal
  - Rajiv Gandhi Cancer Institute & Research Center (RGCIRC), New Delhi
- Italy (18):
  - U.O. di Ematologia e CTMO - Istituti Ospedalieri di Cremona, Cremona, CR
  - IRST - IRCCS U. O. Oncologia Medica, Meldola, FC
  - U.O. Ematologia 1 - IRCCS AOU San Martino-IST, Genova, GE
  - Unita di Ricerca Clinica, Monza, MB
  - Istituto Europeo di Oncologia, Milan, MI
  - Unità semplice di Medicina Nucleare, Latina, NAP
  - Clinica Ematologica - A.O.U. Ospedali Riuniti di Ancona, Torrette Ancona, Palermo
  - Az Ospedaliera Santa Maria, Terni, PG
  - Medicina nucleare, Reggio Emilia, Reggio
  - Radiologia, Reggio Emilia, Reggio
  - SC Ematologia - SC Ematologia - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia, Reggio
  - "Dipartimento di Biotecnologie Cellulari ed Ematologia, Universita ""Sapienza"", Rome, ROME RM
  - IRCSS A.O.U. San Martino - IST - UO Clinica Ematologica, Genova
  - SC Ematologia, Fondazione IRCCS Ist Nazionale dei Tumori, Milan
  - Padiglione 1, Torre delle medicine, 6 piano, Parma
  - Ematologia e Centro Trapianti - AZ Osp. Ospedali Riuniti Marche Nord (AORMN) - Presidio S. Salvatore, Pesaro
  - U.O. Ematologia Universitaria - Dip. Di Oncologia dei Trapianti - AOU Pisana, Pisa
  - Policlinico Universitario Campus Bio- Medico-U.O.C. di Ematologia Trapianto Cellule Staminali, Roma
- Japan (29):
  - East Nagoya Imaging Diagnosis Center, Nagoya, Aichi-ken
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Chiba Cancer Center, Chiba, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Kanazawa Advanced Medical Center, Kanazawa, Ishikawa-ken
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Okocho, Nankoku, Kochi
  - National Hospital Organization Kumamoto Medical Center, Kumamoto, Kumamoto
  - Uozumi Clinic, Kumamoto, Kumamoto
  - Sendai Kousei Hospital, Sendai, Miyagi
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Aizawa Hospital, Matsumoto-shi, Nagano
  - Nagano Red Cross Hospital, Nagano, Nagano
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Hanwa Dai 2 Senboku Hospital, Naka-ku Sakai, Osaka
  - Osaka City University Hospital, Osaka, Osaka
  - Tokushima University Hospital, Tokushima, Tokushima
  - National Hospital Organization Tokyo Medical Center, Meguro-Ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - Yamagata University Hospital, Yamagata, Yamagata
  - Fukuoka Wajiro PET Diagnostic Imaging Clinic, Fukuoka
  - National Hospital Organization Matsumoto Medical Center, Nagano
  - Musashimurayama Hospital, Tokyo
- Lebanon (5):
  - Hammoud Hospital, University Medical Center, Saida, Southern Governate
  - Doctors Center Radiology, Beirut
  - Mount Lebanon Hospital, Beirut
  - Middle East Institute Of Health, El Metn
  - Ain Wazein Hospital, Mount Lebanon
- Mexico (13):
  - Grupo Medico Camino S.C., Mexico City, Mexico City
  - Imagenus, Mexico City, Mexico City
  - Isos Pharmacorp, S.A. de C.V., Mexico City, Mexico City
  - Centro Universitario de Imagen Diagnostica, Radiologia e Imagen del Hospital Universitario, Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Vely Grupo Medico Quirurgico, S.A. de C.V., Cuautitlan Izacalli, State of Mexico
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli, State of Mexico
  - Cirurgia y Ginecobstetricia de Oaxaca, S.A de C.V., Oaxaca City
  - Oaxaca Site Management Organization S.C., Oaxaca City
  - Hospital Angeles Puebla, Puebla City
  - Cancerologia de Queretaro S.C., Querétaro
  - Hospital Infantil Teleton de Oncologia, Querétaro
  - Hospital San Jose Norte, Querétaro
- Peru (3):
  - Instituto Nacional de Enfermedades Neoplasicas, Surquillo, Lima region
  - Pet Scan Peru, Lima
  - Resocentro, Lima
- Philippines (2):
  - University of Philippines Manila-Philippine General Hospital, Manila, National Capital Region
  - St. Luke's Medical Center, Quezon City
- Poland (6):
  - Klinika Nowotworow Ukladu Chlonnego Centrum Onkologii - Instytut im. M. Sklodowskiej-Curie, Warsaw
  - Euromedic Wroclawskie Centrum Medyczne II, Wroclaw
  - Euromedic Wroclawskie Centrum Medyczne III, Wroclaw
  - Dolnoslaskie Centrum Transplantacji Komorkowych z Krajowym Bankiem Dawcow Szpiku, Wroclaw
  - Euromedic Wroclawskie Centrum Medyczne I, Wroclaw
  - Apteka Dolnoslaskiego Centrum Transplantacji Komorkowych z Krajowym Bankiem Dawcow Szpiku, Wroclaw
- Portugal (8):
  - Unidade Local de Saude de Matosinhos E.P.E. - Hospital Pedro Hispano S.A., Matosinhos Municipality, Porto District
  - Hospital de Braga, Braga
  - Hospital CUF Descobertas, Lisbon
  - CIMC, Porto
  - Dr. Campos Costa Clinic, Porto
  - Centro Hospitalar do Porto-Hospital de Santo Antonio E.P.E., Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil E.P.E, Porto
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E., Vila Nova de Gaia
- Puerto Rico (3):
  - Modern Radiology, PSC, Coto Laurel, PR
  - Ad-Vance Medical Research, LLC, Ponce, PR
  - Caribe MRI and CT, Ponce, PR
- Romania (11):
  - Policlinica de Diagnostic Rapid, Hematologie, Brasov
  - Policlinica de Diagnostic Rapid SA, Brasov
  - Spitalul Clinic Colentina, Bucharest
  - Hiperdia Ritmului, Bucharest
  - Affidea Fundeni, Bucharest
  - Affidea Romania SRL, Bucharest
  - Spitalul Clinic Coltea, Clinica de Hematologie, Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Laborator Radiologie si Imagistica Medicala, Cluj-Napoca
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Sectia Oncologie Medicala, Cluj-Napoca
  - Clinica de Hematologie-Institutul Oncologic, Prof. Dr. Ion Chiricuta, Cluj-Napoca
  - CT Clinic S.R.L., Cluj-Napoca
- Russia (31):
  - A.Tsyb Medical Radiological Research Centre -, Obninsk, Kaluga Oblast
  - State Healthcare Institution Republican Oncology Dispensary, Saransk, Mordovian Republic
  - "SBHI of NNR ""Nizhniy Novgorod Regional Clinical Hospital n.a. N.A. Semashko""", Nizhny Novgorod, Nizhniy Novgorod Region
  - LLC MC "MRT-Diagnostika", Nizhny Novgorod, Nizhniy Novgorod Region
  - FSBI "Russian Research Centre of Radiology and Surgical Technologies" of MoH of RF, Saint Petersburg, Pesochniy TOWN
  - FSBI "Russian Research Centre of Radiology and Surgical Technologies", Saint Petersburg, Pesochniy TOWN
  - FSBI "Russian Research Centre of Radiology and Surgical Technologies, Saint Petersburg, Pesochniy TOWN
  - FSBI 'Russian Research Centre of Radiology and Surgical Technologies, Saint Petersburg, Pesochniy TOWN
  - FSBI "Russian Research Centre of Radiology and Surgical Technologies n.a. A.M. Granov" of MoH of RF, Saint Petersburg, Pesochniy
  - FSBI "Russian Research Centre of Radiology and Surgical Technologies named after academician, Saint Petersburg, Pesochniy
  - FSBI "Russian Research Centre of Radiology and Surgical Technologies, Saint Petersburg, Pesochniy
  - FSBI 'National Medical Oncology Research Centre n.a. N.N.Petrov', Saint Petersburg, Pos.pesochny
  - Branch office of LLC 'PET-Technology' at Ufa city, Ufa, Republic Bashkortostan
  - State Budgetary Healthcare Institution "Republican Clinical Oncology Dispensary of the Ministry, Ufa, Republic Bashkortostan
  - FSBI "Russian Research Centre of Radiology and Surgical Technologies" of MoH of RF, Pesochniy Town, Sankt-Peterburg
  - Private medical institution "Euromedservice", Pushkin, Sankt-Peterburg
  - Federal State-Financed Institution 'North-Caucasian Research and Clinical Center', Lermontov, Stavropol Kray
  - SBHI of Stavropol Region "Pyatigorsk Interdistrict Oncology Dispensary, Pyatigorsk, Stavropol Kray
  - "State Budget Healthcare Institution ""Chelyabinsk Regional Clinical Center of Oncology, Chelyabinsk
  - FSBSI 'N.N.Blokhin Russian Cancer Research Center' of MoH of RF, Moscow
  - Russian Cancer Research Centre them N.N. Blokhin, Moscow
  - LLC "VitaMed", Moscow
  - SBHI of Moscow City Clinical Hospital n.a. S.P.Botkin of Healthcare Department of Moscow, Moscow
  - Ramsay Diagnostics, Moscow
  - Dr. Berezin Medical Institute, Saint Petersburg
  - State Budgetary Institution of Healthcare "Leningrad Regional Clinical Hospital", Saint Petersburg
  - N.P. Bechtereva Institute of Human Brain of the Russian Academy of Sciences, Saint Petersburg
  - N.P. Bechtereva Institute of the Human Brain of the Russian Academy of Sciences, Saint Petersburg
  - Non-state healthcare institution "Road Clinical Hospital of Joint Stock Company "Russian Railways", Saint-Petersurg
  - Yaroslavl State Medical Academy, Yaroslavl
  - GBUZ of Yaroslavl Region "Regional Clinical Hospital", Yaroslavl
- South Africa (8):
  - NIKSCH & PARTNERS t/a CAPITAL RADIOLOGY, Groenkloof, Gauteng
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Department of Medical Oncology, University of Pretoria, Steve Biko Academic Hospitals Complex, Pretoria, Gauteng
  - Albert Alberts Stem Cell Transplant Centre, Pretoria, Gauteng
  - Dr JN De Jong and Partners t/a East Rad, Pretoria, Gauteng
  - NIKSCH & PARTNERS t/a CAPITAL RADIOLOGY, Pretoria, Gauteng
  - Drs Sulman & Partners Specialist Radiologists, Rosebank, Gauteng
  - Drs Bloch & Partners Incorporated, Sandton, Gauteng
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Ulsan University Hospital, Ulsan, Korea
  - Inje University Busan Paik Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (23):
  - Hospital Parc Tauli, Sabadell, Barcelona
  - Onkologikoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario Sanitas La Zarzuela, Aravaca, Madrid
  - Hospital Rey Juan Carlos, Móstoles, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital do Meixoeiro Complejo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Modelo, A Coruña
  - Hospital Del Mar, Barcelona
  - Hospital Quiron de Barcelona, IEC, Barcelona
  - CETIR, Centre Medic, Barcelona
  - Radiodiagnostic CETIR - Clinica del Pilar, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Sanitas La Moraleja, Madrid
  - Centro CIMES, Málaga
  - Hospital universitario Virgen de la Victoria, Málaga
  - Centro Mario Gallegos, Málaga
  - Complejo Hospitalario de Ourense. Hematología, Ourense
  - Hospital Universitario Virgen del Rocio, Seville
  - H. Quiron Zaragoza, Zaragoza
  - Hospital de Dia Quiron Zaragoza, Zaragoza
- Switzerland (6):
  - Universitatsspital Basel, Basel
  - Inselspital Bern, Bern
  - Apotheke, Spital STS AG, Thun
  - Onkologiezentrum Thun-Berner Oberland Spital Sts Ag, Thun
  - Kantonsapotheke Zuerich, Zurich
  - UniversitaetsSpital Zuerich, Zurich
- Thailand (3):
  - Cardiology Unit,Department of Medicine, Faculty of Medicine, Ramathibodi Hospital,, Bangkok
  - Department of Radiology, Ramathibodi Hospital, Bangkok
  - National Cancer Institute, Bangkok
- Turkey (Türkiye) (17):
  - Hacettepe Universitesi Tip Fakultesi Onkoloji Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Eg. ve Aras., Ankara
  - Ultramar Tibbi Gorunteleme Merkezi, Ankara
  - Ultramar Tibbi Goruntuleme Merkezi, Ankara
  - Integra Gurses Teshis Tedavi ve Saglik Hizmetleri A.S., Ankara
  - Adnan Menderes University Medical Faculty, Aydin
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama, Gaziantep
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Ic Hastaliklari Anabilim Dali, Izmir
  - EGE-RAD Bilgisayarli Tomografi Ozel Saglik Hizmetleri ve Malzemeleri Tic.Ltd.Sti., Izmir
  - Erciyes Universitesi Tip Fakultesi Nukleer Tip Laboratuvari, Kayseri
  - Erciyes Universitesi Tip Fakultesi Radyoloji Laboratuvari, Kayseri
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Inonu Universitesi Tip Fakultesi Turgut Ozal Tip Merkezi, Malatya
  - Celal Bayar University Medical Faculty, Manisa
  - Ondokuz Mayis Universitesi Tip Fakultesi, Samsun
- Ukraine (11):
  - "MedX-Ray International Group" LLC, Obukhiv, Kyiv Oblast
  - "Mediks-rey International Group" LLC, Obukhiv District, Kyiv Oblast
  - "MedX-rey International Group" LLC, Obukhiv District, Kyiv Oblast
  - "Municipal Institution ""Chernivtsi Regional Clinical Oncology Center"",, Chernivtsi
  - MI 'City Dnipropetrovsk Multi-field Clin. Hospital #4 of DRC',, Dnipropetrovsk
  - Municipal Non-Profit Enterprise "Regional Oncology Centre", Kharkiv
  - National Cancer Institute, Kyiv
  - "Central City Clinical Hospital, City Oncology Center, SHEI ""Uzhhorod National University"", Chair, Uzhhorod
  - Podilskyy Regional Oncology Center, Chemotherapy Department, Vinnytsia
  - Municipal Establishment 'Zaporizhzhia Regional Clinical Oncology Dispensary', Zaporizhzhia
  - LLC "Diaservis", Zaporizhzhia
- United Kingdom (7):
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, Essex
  - Cobalt Diagnostic Imaging, Cheltenham, Glos.
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Barts Health NHS Trust, London
  - Positron Emission Tomography (PET) Centre, Newcastle upon Tyne
  - City Hospitals Sunderland NHS Foundation Trust-Sunderland Royal Hospital, Sunderland
  - Diagnostic Imaging, Sunderland

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Courville J, Nastoupil L, Kaila N, Kelton J, Zhang J, Alcasid A, Nava-Parada P. Factors Influencing Infusion-Related Reactions Following Dosing of Reference Rituximab and PF-05280586, a Rituximab Biosimilar. BioDrugs. 2021 Jul;35(4):459-468. doi: 10.1007/s40259-021-00487-6. Epub 2021 Jun 21. PMID 34152584
- [Derived] Sharman JP, Liberati AM, Ishizawa K, Khan T, Robbins J, Alcasid A, Rosenberg JA, Aurer I. A Randomized, Double-Blind, Efficacy and Safety Study of PF-05280586 (a Rituximab Biosimilar) Compared with Rituximab Reference Product (MabThera(R)) in Subjects with Previously Untreated CD20-Positive, Low-Tumor-Burden Follicular Lymphoma (LTB-FL). BioDrugs. 2020 Apr;34(2):171-181. doi: 10.1007/s40259-019-00398-7. PMID 31820339
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3281006

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 394 participants were enrolled and randomized in 1:1 ratio to 1 of the 2 study treatment arms: PF-05280586 (Rituximab-Pfizer) and Rituximab-EU (MabThera®).
Groups:
- Rituximab-EU: Participants received Rituximab-EU intravenous (IV) infusion at a dose of 375 milligrams per meter square (mg/m^2) on Day 1, 8, 15, and 22. The maximum dose that could be infused in 1 day was 1125 mg.
- PF-05280586: Participants received PF-05280586 IV infusion at a dose of 375 mg/m^2 on Day 1, 8, 15, and 22. The maximum dose that could be infused in 1 day was 1125 mg.
Period: Overall Study
Arm/Group | Rituximab-EU | PF-05280586
Started | 198 | 196
Treated | 197 | 196
Completed | 170 | 170
Not Completed | 28 | 26
Not completed — Insufficient clinical response | 4 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — No longer willing to participate | 3 | 4
Not completed — Progressive disease | 20 | 14
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab-EU | PF-05280586 | Total
Number analyzed (Participants) | 198 | 196 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (12.8) | 58.7 (12.1) | 58.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 110 | 216
  Male | 92 | 86 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 31 | 57
  Not Hispanic or Latino | 172 | 165 | 337
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 44 | 30 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 146 | 158 | 304
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR): Percentage of Participants With Overall Response (OR) at Week 26
Description: ORR was defined as the percentage of participants who achieved complete response (CR) or partial response (PR) in accordance with the revised response criteria for malignant lymphoma (Cheson 2007). CR was defined as disappearance of all evidence of disease. PR was defined as regression of measureable disease and no new sites.
Time Frame: Week 26
Population: ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 198 | 196
percentage of participants | 70.7 [63.8 to 76.9] | 75.5 [68.9 to 81.4]
Statistical Analysis 1: Comparison: Rituximab-EU vs PF-05280586; Difference in ORR between PF-05280586 and rituximab-EU was computed using the stratified Mantel-Haenszel method. The 95% confidence interval for the difference was calculated using the asymptotic stratified method proposed by Miettinen and Nurminen; Test type: Equivalence — Equivalence was tested within the pre-specified margins of (-16%, 16%) 95% confidence interval; Difference in ORR = 4.66, 95% CI 2-sided [-4.16 to 13.47]

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in participants who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events after first dose of study drug that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious.
Time Frame: Baseline up to Week 52
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 196
Participants
  AEs | 145 | 156
  SAEs | 15 | 17

3. Secondary Outcome: Number of Participants With Treatment Related Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events after first dose of study drug that were absent before treatment or that worsened relative to pretreatment state. Relatedness to treatment was assessed by investigator. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to Week 52
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 196
Participants
  AEs | 94 | 86
  SAEs | 2 | 2

4. Secondary Outcome: Number of Participants With Grade 3 or Higher Treatment-Emergent Adverse Events (AEs) as Graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03
Description: An AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. Grade 1=Mild, asymptomatic or mild symptoms, Grade 2=Moderate; minimal, local or noninvasive intervention indicated, Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life threatening) events caused participant to be in imminent danger of death. Grade 5 = death. Treatment-emergent were events after first dose of study drug that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Week 52
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 196
Participants | 26 | 28

5. Secondary Outcome: Number of Participants With Grade 3 or Higher Treatment-Related Treatment-Emergent Adverse Events (AEs) as Graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Grade 1=Mild, asymptomatic or mild symptoms, Grade 2=Moderate; minimal, local or noninvasive intervention indicated; Grade 3 (Severe) events=unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 (Life-threatening) events caused participant to be in imminent danger of death. Grade 5 = death. Treatment-emergent were events after first dose of study drug that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Week 52
Population: Safety population included all participants who received at least 1 dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 196
Participants | 8 | 9

6. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Criteria for clinically significant laboratory abnormalities included total bilirubin (TB) less than (<) 2*upper limit of normal (ULN), alanine aminotransferase (ALT)<3*ULN; TB<2*ULN, ALT more than (>) 3 equal to (=) *ULN; TB<2*ULN, aspartate aminotransferase (AST)<3*ULN; TB<2*ULN, AST>=3*ULN. Data for only those categories are reported for which at least one participant had clinically significant laboratory abnormality.
Time Frame: Baseline up to Week 52
Population: Safety population included all participants who received at least 1 dose of any study drug. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 195
Participants
  TB<2*ULN, ALT<3*ULN | 194 | 192
  TB<2*ULN, ALT>=3*ULN | 3 | 3
  TB<2*ULN, AST<3*ULN | 196 | 195
  TB<2*ULN, AST>=3*ULN | 1 | 0

7. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time (in months) from date of randomization to first progression of disease based on central review, death due to any cause, or permanent discontinuation from treatment, or discontinuation from study for any reason, whichever came first. Progression was defined as any new lesion or increase by greater than or equal to (>=) 50% of previously involved sites from nadir. TTF was calculated using Kaplan-Meier method.
Time Frame: From randomization until disease progression, death or permanent discontinuation from treatment/study due to any reason, or up to Week 52
Population: ITT population included all participants who were randomized. Here. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 48 | 54
months | 18.9 [12.6 to 18.9] | NA [12.3 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated.
Statistical Analysis 1: Comparison: Rituximab-EU vs PF-05280586; Test type: Superiority; p = 0.450, Log Rank — A log-rank test stratified by follicular lymphoma international prognostic index 2 (FLIPI2) risk was used to compare the treatment groups with respect to TTF at a 2-sided alpha level of 0.05; Hazard Ratio (HR) = 1.163, 95% CI 2-sided [0.786 to 1.720] — Hazard ratio and its confidence intervals (CIs) were estimated from Cox Proportional hazards model stratified by FLIPI2 risk categorization

8. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time (in months) from date of randomization to first progression of disease (PD) based on central review or death due to any cause in the absence of documented PD. PD was defined as any new lesion or increase by >=50% of previously involved sites from nadir. PFS was calculated using Kaplan-Meier method.
Time Frame: From randomization until disease progression or death due to any cause or up to Week 52
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 28 | 37
months | 18.9 [12.6 to 18.9] | NA [NA to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated.
Statistical Analysis 1: Comparison: Rituximab-EU vs PF-05280586; Test type: Superiority; p = 0.189, Log Rank; A log-rank test stratified by FLIPI2 risk was used to compare the treatment groups with respect to PFS at a 2-sided alpha level of 0.05; Hazard Ratio (HR) = 1.393, 95% CI 2-sided [0.847 to 2.291] — Hazard ratio and its CIs were estimated from Cox Proportional hazards model stratified by FLIPI2 risk categorization

9. Secondary Outcome: Percentage of Participants With Complete Remission (CR) at Week 26
Description: Complete Remission (CR) was defined as disappearance of all evidence of disease. CR was assessed by central review based on scans done at Week 26.
Time Frame: Week 26
Population: ITT population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 198 | 196
percentage of participants | 28.3 [22.1 to 35.1] | 26.0 [20.0 to 32.8]
Statistical Analysis 1: Comparison: Rituximab-EU vs PF-05280586; Difference in CR between PF-05280586 and rituximab-EU was computed using the stratified Mantel-Haenszel method. The 95% confidence interval for the difference was calculated using the asymptotic stratified method proposed by Miettinen and Nurminen; Test type: Superiority; Mean Difference (Final Values) = -2.31, 95% CI 2-sided [-11.09 to 6.50]

10. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time (in months) from date of the first documentation of overall response (CR or PR) to the first documentation of progressive disease (PD) based on central review or to death due to any cause in the absence of documented PD. CR was defined as disappearance of all evidence of disease. PR was defined as regression of measureable disease and no new sites. PD was defined as any new lesion or increase by >=50% of previously involved sites from nadir. DOR was calculated using Kaplan-Meier method.
Time Frame: From date of first documentation of overall response to first documentation of PD or to death due to any cause in absence of PD or up to Week 52
Population: The response-evaluable population was defined as all randomized participants who received at least 1 dose of study drug, had adequate disease assessment at baseline, and at least 1 post baseline response assessment. Here. 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 19 | 28
months | 15.4 [10.4 to 15.4] | NA [9.6 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated.
Statistical Analysis 1: Comparison: Rituximab-EU vs PF-05280586; Test type: Superiority; p = 0.185, Log Rank — A log-rank test stratified by FLIPI2 risk was used to compare the treatment groups with respect to DOR at a 2-sided alpha level of 0.05; Hazard Ratio (HR) = 1.492, 95% CI 2-sided [0.823 to 2.704] — Hazard ratio and its CIs were estimated from Cox Proportional hazards model stratified by FLIPI2 risk categorization

11. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time (in months) from date of randomization to death due to any cause. For participants who were alive, overall survival was censored at the last contact. Overall survival was calculated using Kaplan-Meier method.
Time Frame: From randomization until death due to any cause or up to Week 52
Population: ITT population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 198 | 196
months | 18.9 [NA to NA] — Due to single participant with an event, lower and upper limit of 95% CI could not be calculated. | NA [NA to NA] — Due to single participant with an event, median, lower and upper limit of 95% CI could not be calculated.
Statistical Analysis 1: Comparison: Rituximab-EU vs PF-05280586; Test type: Superiority; p = 0.319, Log Rank — A log-rank test stratified by FLIPI2 risk was used to compare the treatment groups with respect to overall survival at a 2-sided alpha level of 0.05; Hazard Ratio (HR) = 2.94, 95% CI 2-sided [lower limit 0.000] (Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated.) — Hazard ratio and its CIs were estimated from Cox Proportional hazards model stratified by FLIPI2 risk categorization

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-05280586 and Rituximab-EU
Time Frame: Predose (within 4 hours prior to start of infusion) on Days 1, 8, 15 and 22; within 15 minutes prior to end of infusion on Days 1 and 22
Population: The pharmacokinetic analysis set (PKAS) included participants who received at least 1 dose of any study drug and who provided at least one post-dose pharmacokinetic concentration. Here, 'Overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 132 | 138
nanograms per milliliter (ng/mL) | 334848.88 (33) | 337708.05 (36)

13. Secondary Outcome: Minimum Observed (Trough) Serum Concentration (Ctrough) of PF-05280586 and Rituximab-EU
Time Frame: Predose (within 4 hours prior to the start of dosing) on Day 1, 8, 15, and 22
Population: The pharmacokinetic analysis set (PKAS) included participants who received at least 1 dose of any study drug and who provided at least one post-dose pharmacokinetic concentration. Here 'Number analyzed' signifies number of participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 196
ng/mL
  Day 1: number analyzed (Participants) | 195 | 192
  Day 1 | 0.01 (577) | 0.01 (1320)
  Day 8: number analyzed (Participants) | 197 | 194
  Day 8 | 62311.74 (47) | 66669.15 (45)
  Day 15: number analyzed (Participants) | 194 | 193
  Day 15 | 109619.73 (43) | 119026.91 (29)
  Day 22: number analyzed (Participants) | 194 | 194
  Day 22 | 144650.79 (68) | 158294.91 (32)

14. Secondary Outcome: Cluster of Differentiation (CD) 19-Positive B-Cell Counts
Time Frame: Baseline, Week 2, 3, 4, 5, 13, 26, 39, 52
Population: The modified ITT (mITT) Population included all participants who were randomized and received at least 1 dose of any study drug. Here 'Number analyzed' signifies number of participants evaluable for this outcome measure at specified time points.
Measure: Median (Full Range); unit: Cells per microliter
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 196
Cells per microliter
  Baseline: number analyzed (Participants) | 173 | 175
  Baseline | 114.2 [0.6 to 2313.1] | 119.9 [10.9 to 1310.1]
  Week 2: number analyzed (Participants) | 168 | 159
  Week 2 | 1.0 [0.2 to 44.8] | 0.8 [0.2 to 136.0]
  Week 3: number analyzed (Participants) | 149 | 149
  Week 3 | 0.6 [0.2 to 19.5] | 0.6 [0.2 to 248.1]
  Week 4: number analyzed (Participants) | 143 | 114
  Week 4 | 0.5 [0.2 to 8.7] | 0.4 [0.2 to 144.5]
  Week 5: number analyzed (Participants) | 118 | 128
  Week 5 | 0.5 [0.2 to 19.0] | 0.4 [0.2 to 19.0]
  Week 13: number analyzed (Participants) | 106 | 103
  Week 13 | 0.5 [0.2 to 130.7] | 0.5 [0.2 to 183.7]
  Week 26: number analyzed (Participants) | 142 | 123
  Week 26 | 1.2 [0.2 to 496.5] | 0.9 [0.2 to 329.8]
  Week 39: number analyzed (Participants) | 157 | 135
  Week 39 | 21.7 [0.3 to 341.0] | 10.7 [0.2 to 442.7]
  Week 52: number analyzed (Participants) | 151 | 147
  Week 52 | 60.8 [1.4 to 413.0] | 51.6 [0.3 to 597.9]

15. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADAs) and Neutralizing Antibodies (NAbs)
Description: Human serum ADA samples were analyzed for the presence or absence of anti-rituximab antibodies or anti-PF-05280586 antibodies using the validated drug-specific assay with a tiered approach using screening, confirmation and titer/quantitation. Human NAb serum samples testing ADA positive were analyzed for the presence or absence of neutralizing anti-rituximab antibody and neutralizing anti-PF-05280586 antibody using the validated drug-specific assay with a tiered approach using screening, confirmation and titer/quantitation. Participants with their ADA titer >= 1.88 were considered to be ADA positive. Only participants with a positive ADA result were further tested for NAb.
Time Frame: Baseline up to Week 52
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 195
Participants
  ADA Positive | 39 | 43
  NAB Positive: number analyzed (Participants) | 39 | 43
  NAB Positive | 0 | 0

16. Secondary Outcome: Number of Participants Reporting Immune-Based Adverse Effects
Description: Immune-based adverse effects included infusion related reaction (IRR), adverse events which fulfill Sampson's criteria, and adverse events which belong to the Standardized Medical Dictionary for Regulatory Activities (MedDRA) Queries (SMQs) anaphylaxis or hypersensitivity reactions. Potential allergic and anaphylactic reactions were identified programmatically based on the criteria of Sampson et al, (2006).
Time Frame: Baseline up to Week 52
Population: The Safety analysis population include all participants who received at least 1 dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab-EU | PF-05280586
Number analyzed (Participants) | 197 | 196
Participants
  IRR reported | 59 | 49
  AE based on Sampson's criteria | 17 | 17
  Anaphylaxis/Hypersensitivity (SMQ) | 48 | 39

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (up to 52 weeks)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis was performed on safety population.
Arm/Group | Rituximab-EU | PF-05280586
All-Cause Mortality (participants affected / at risk) | 1/197 | 1/196
Serious Adverse Events (participants affected / at risk) | 15/197 | 17/196
Other Adverse Events (participants affected / at risk) | 143/197 | 153/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab-EU (N=197) | PF-05280586 (N=196)
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 1
Disease progression (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Serum sickness (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral sinusitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Rituximab-EU (N=197) | PF-05280586 (N=196)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 5
Sinus bradycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 2
Ear disorder (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1
Ear pruritus (Ear and labyrinth disorders) | 2 | 3
Hypoacusis (Ear and labyrinth disorders) | 2 | 2
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Thyroid cyst (Endocrine disorders) | 0 | 1
Accommodation disorder (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 2
Conjunctival disorder (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 2 | 0
Erythema of eyelid (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 3 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Meibomianitis (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 7
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 9
Asthenia (General disorders) | 13 | 9
Axillary pain (General disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Catheter site pain (General disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 8 | 8
Catheter site related reaction (General disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 12 | 14
Chest discomfort (General disorders) | 1 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 0
Discomfort (General disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Faeces soft (Gastrointestinal disorders) | 1 | 0
Face oedema (General disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 3
Fatigue (General disorders) | 13 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Feeling cold (General disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Feeling hot (General disorders) | 2 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Lip oedema (Gastrointestinal disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 2
Mouth swelling (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 17 | 15
Odynophagia (Gastrointestinal disorders) | 1 | 1
Oral discomfort (Gastrointestinal disorders) | 0 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1
Influenza like illness (General disorders) | 4 | 2
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Salivary gland pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0
Infusion site bruising (General disorders) | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 7 | 3
General physical health deterioration (General disorders) | 1 | 0
Infusion site erythema (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Infusion site pain (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 3
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 7 | 2
Pain (General disorders) | 3 | 3
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 11 | 11
Suprapubic pain (General disorders) | 1 | 0
Swelling (General disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 1 | 2
Cytokine release syndrome (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 1
Atypical mycobacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 7 | 3
Cellulitis (Infections and infestations) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Conjunctivitis (Infections and infestations) | 3 | 0
Cystitis (Infections and infestations) | 3 | 1
Chest injury (Injury, poisoning and procedural complications) | 1 | 1
Cystitis bacterial (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 2
Genital herpes (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 1
Infected bite (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 6 | 4
Laryngitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 9 | 5
Oral herpes (Infections and infestations) | 2 | 3
Otitis externa fungal (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Pertussis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 4 | 4
Pneumonia (Infections and infestations) | 0 | 1
Purulence (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 3
Rhinitis (Infections and infestations) | 3 | 1
Sinusitis (Infections and infestations) | 2 | 5
Skin infection (Infections and infestations) | 2 | 0
Sycosis barbae (Infections and infestations) | 1 | 0
Systemic infection (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Trichophytosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 9
Urinary tract infection (Infections and infestations) | 5 | 4
Viral infection (Infections and infestations) | 0 | 1
Viral pharyngitis (Infections and infestations) | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 5
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 58 | 49
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Neck injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 3
Blood potassium increased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 1 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 5
Neutrophil count increased (Investigations) | 1 | 0
Serum ferritin decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 4
Breath sounds abnormal (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 8
Bone loss (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 7
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 | 0
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 6 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 19 | 16
Hypoaesthesia (Nervous system disorders) | 1 | 1
Hypotonia (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 3 | 2
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 3
Somnolence (Nervous system disorders) | 3 | 2
Speech disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 7 | 6
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 3
Gastrointestinal somatic symptom disorder (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 8 | 5
Irritability (Psychiatric disorders) | 1 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 2
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 1 | 0
Strangury (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1
Genital burning sensation (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 3
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 7
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Menopause (Social circumstances) | 0/106 | 1/110
Deep vein thrombosis (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 4 | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 10
Hypertension (Vascular disorders) | 7 | 5
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 2
Scab (Skin and subcutaneous tissue disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 6 | 3
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 13
Entropion (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-04-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT02213263/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT02213263/SAP_001.pdf